CLINICAL TRIAL: NCT01271036
Title: A Single-Center, Medically Supervised, Safety Evaluation Study of a Sensitive Sensual Touch and Personal Lubricant Product in Couples
Brief Title: Safety Study of a Sensitive Sensual Touch and Personal Lubricant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Healthcare Products Division of McNEIL-PPC, Inc. (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: KOYNAP0010
Record Dates: First submitted 2011-01-04; First posted 2011-01-06 (Estimated); Results first posted 2014-03-04 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2013-09

CONDITIONS: Inadequate Lubrication
Keywords: Lubricating Agents; Personal Lubricant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Formula PD-F-7716 (Experimental): Apply a dime-size amount on each application site as instructed during the 1-week study period
  Interventions: Device: Formula PD-F-7716

INTERVENTIONS:
Device: Formula PD-F-7716 — Apply a dime-size amount on each application site as instructed during the 1-week study period
  Other Names: KY BRAND TOUCH® 2-in-1; Sensitive Massage Lotion and Personal Lubricant

SUMMARY:
This is a one week study designed to test the safety of a personal lubricant during in-home use for subjects who perceive themselves as having sensitive skin.

DETAILED DESCRIPTION:
This is a single-center, medically supervised, single-arm study to evaluate the safety of an all over 2-in-1 sensual touch lotion and personal lubricant product in home-use conditions via clinical assessment. The study will consist of two visits. Subjects who meet the entrance criteria will receive investigational product (IP) and four subjective questionnaires for at-home completion. The subjects will be required to use the IP at least two times on each application site, as instructed over the 1-week home-use period. At the end of the study (Visit 2) subjects will return to the study site, at which time all unused IP and questionnaires will be returned and a final clinical assessment will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Normal, healthy adults in a stable, monogamous, ongoing heterosexual relationship with current partner for at least 6 months
* Subjects comfortable discussing sensitive topics such as personal hygiene, menstruation and sexuality
* At least one partner in the couple has sensitive skin per protocol-defined criteria
* Able to read and understand English
* Voluntarily signs an Informed Consent document after the trial has been explained
* Willing to follow all study procedures, including birth control requirements

Exclusion Criteria:

* Any medical or mental health history or condition, or use of any product, drug or medication that per protocol (or in the opinion of the Investigator) might compromise the participant's safety or the analysis of results
* Participation as a research subject within timelines dictated by protocol
* Participants with relationships or employment outside protocol-defined parameters

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2010-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherryl Frisch, Study Director — Johnson & Johnson Consumer and Personal Products Worldwide
Locations (1):
- Thomas J Stephens & Associates, Inc., Colorado Springs, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only one IP was used per couple in this single-arm study. At baseline (visit 1), all qualified subjects received the IP for use per protocol.
Groups:
- Males: Male Participants (K-Y Brand TOUCH 2-in-1)
- Female: Female Participants (K-Y Brand TOUCH 2-in-1)
Period: Overall Study
Arm/Group | Males | Female
Started | 62 | 62
Completed | 62 | 62
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- Male: Male Participants
- Female: Female Participants
- Total: Total of all reporting groups
Arm/Group | Male | Female | Total
Number analyzed (Participants) | 62 | 62 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (13.8) | 42.0 (12.7) | 42.8 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 62 | 62
  Male | 62 | 0 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 62 | 62 | 124
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 5 | 13
  White | 51 | 53 | 104
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 62 | 62 | 124
Menopausal Status [Number; unit: Participants]
  Premenopausal | NA — Data Not Available because menopausal status is not applicable to male subjects. | 46 | 46
  Postmenopausal | NA — Data Not Available because menopausal status is not applicable to male subjects. | 16 | 16
Total Couples with Sensitive Skin [Number; unit: participants]
  Couple with Male Partner with Sensitive Skin | 3 | 0 | 3
  Couple with Female Partner with Sensitive Skin | 0 | 46 | 46
  Couple with Both Partners with Sensitive Skin | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Physical Irritation Scores
Description: Severity of physical irritation scored by the Investigator on a scale from 0 (no irritation) to 6 (presence of lesions). Since a score of 0 is required at baseline for inclusion in the study, this any score represents a change from baseline and the trial is considered baseline-controlled. The number of participants with physical irritation scores after one week was recorded (along with categorical severity).
Time Frame: One week
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Male | Female
Number analyzed (Participants) | 62 | 62
Participants
  No Irritation, Either Region | 61 | 61
  Mild Irritation, Neck Region | 1 | 0
  Mild Irritation, Genital Region | 0 | 1

2. Secondary Outcome: Number of Participants Reporting Subjective Irritation - Genital Application 1
Description: Participants were asked to rate specific sensations they experienced during each application at each site (genital and neck) on a five-point categorical severity scale from mild to excruciating. The sensations included itching, burning, stinging, tingling, warming, and cooling. The number of participants with subjective irritation scores after one week was recorded.
Time Frame: One week
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Male | Female
Number analyzed (Participants) | 62 | 62
Participants
  Baseline | 0 | 0
  Itching | 4 | 3
  Burning | 1 | 6
  Stinging | 1 | 2
  Tingling | 7 | 13
  Warming | 15 | 22
  Cooling | 12 | 13

3. Secondary Outcome: Number of Participants Reporting Subjective Irritation - Genital Application 2
Description: as for outcome 2
Time Frame: One week
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Male | Female
Number analyzed (Participants) | 62 | 62
Participants
  Baseline | 0 | 0
  Itching | 2 | 1
  Burning | 1 | 5
  Stinging | 1 | 1
  Tingling | 5 | 10
  Warming | 17 | 18
  Cooling | 12 | 10

4. Secondary Outcome: Number of Participants Reporting Subjective Irritation - Neck Application 1
Description: as for outcome 2
Time Frame: One week
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Male | Female
Number analyzed (Participants) | 62 | 62
Participants
  Baseline | 0 | 0
  Itching | 1 | 2
  Burning | 1 | 0
  Stinging | 2 | 1
  Tingling | 4 | 8
  Warming | 10 | 13
  Cooling | 14 | 15

5. Secondary Outcome: Number of Participants Reporting Subjective Irritation - Neck Application 2
Description: as for outcome 2
Time Frame: One week
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Male | Female
Number analyzed (Participants) | 62 | 62
Participants
  Baseline | 0 | 0
  Itching | 2 | 4
  Burning | 1 | 0
  Stinging | 1 | 0
  Tingling | 1 | 9
  Warming | 10 | 12
  Cooling | 16 | 15

ADVERSE EVENTS:
Time Frame: 1 Week (+30 days for Serious Adverse Events, and beyond if assessed as possibly treatment related)
Description: Adverse Events were collected from all study subjects via subjective questionnaire and physical examination. Participants are counted one time for each adverse event they experienced.
Arm/Group | Male | Female
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/62
Other Adverse Events (participants affected / at risk) | 7/62 | 17/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Male (N=62) | Female (N=62)
Application Site Pain (e.g., burning, stinging) (General disorders) | 2 | 8
Application Site Pruritus (e.g., itching) (General disorders) | 4 | 6
Application Site Erythema (General disorders) | 1 | 2
Application Site Excoriation (General disorders) | 0 | 2
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ankle Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study is considered a work made for hire and the Sponsor retains all rights to publish results.